CLINICAL TRIAL: NCT00010621
Title: Complementary Medicine Approaches to TMD Pain Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: P50AT000076-01P1 (NIH); P50AT000076-01 (NIH); NCT00009334 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Acupuncture Therapy; Musculoskeletal Manipulations

INTERVENTIONS:
Procedure: Acupuncture
Procedure: chiropractic therapy
Procedure: bodywork therapy

SUMMARY:
This study will determine whether selected complementary approaches to temporomandibular joint (TMJ) pain management-acupuncture are as effective as usual care.

DETAILED DESCRIPTION:
Temporomandibular disorders are characterized by pain and tenderness in the muscles of mastication and/or the (TMJ), limitations of jaw opening often accompanied by deviations in mandibular path, and clicking, popping or grating TMJ sounds. This study will compare the effectiveness of the complementary therapies chiropractic therapy and bodywork therapy to the standard of care for TMJ pain. If these complementary interventions are shown to be effective, the goal is to design and implement a Phase III clinical trial to further evaluate the health consequences and cost of these therapies.

Participants will be evaluated at baseline, and 6 and 12 months post-intervention. Clinical examinations, saliva samples to assess salivary cortisol levels, and a series of questionnaires to assess pain and grade of dysfunctional pain, psychological functioning, and other physical symptoms will be used to assess outcomes. The investigators will passively monitor health care utilization within KPNW using clinical, research, and administrative databases.

ELIGIBILITY:
Inclusion Criteria:

* Psychologically functional TMD patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Alex White, Principal Investigator — Center for Health Research (CHR), Kaiser Foundation Hospitals
Locations (1):
- Center for Health Research, Portland, Oregon, United States